CLINICAL TRIAL: NCT00382447
Title: Breath Actuated Nebulizer Study Protocol
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to put forth the human resources for patient enrollment
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CCC# 26168
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
Keywords: breath actuated nebulizer; nebulizer
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Standard nebulizer versus standard breath actuated nebulizer
  Interventions: Device: standard nebulizer; Device: breath actuated nebulizer

INTERVENTIONS:
Device: standard nebulizer — Standard small volume nebulizer for aerosolized medication delivery
Device: breath actuated nebulizer — Nebulizer that dispenses medication only during the inspiratory phase

SUMMARY:
Comparison of the researchers' standard nebulizer and a breath actuated nebulizer to examine if breathing medication can be delivered more quickly and as effectively or more effectively than the standard nebulizer.

DETAILED DESCRIPTION:
Background:

Generic nebulizers as well as breath actuated nebulizers have been available and FDA approved to administer therapy for years. Recently there has been interest in using breath actuated nebulizers to stream-line patient care in the hospital setting. Literature has found that breath actuated nebulizers are not only faster at delivering an equivalent dose, but more effective when measuring patient response to that therapy. There is no standard for method of converting from generic nebulizers to breath actuated technology.

Objectives:

We want to evaluate the use of Breath Actuated Nebulizer (BAN) technology versus generic nebulizers to improve quality of patient treatments and reduce nebulization duration to allow staff time to do complete patient assessments.

Inclusion Criteria:

* Adult patients with orders for routine 2.5 mg albuterol sulfate nebulizer therapy ordered either Q4 or Q6 hours who consent to the study.

Exclusion Criteria:

* Adults with nebulizer therapy ordered more frequently than Q4 hours.
* Adults with nebulizer therapy ordered less frequently than Q6 hours.
* Pregnant patients are excluded.
* Adults with orders for albuterol sulfate > 2.5 mg.
* Adults in the intensive care unit (ICU) or Emergency Department.

Protocol:

1. Adult patient ordered for Q4 to Q6 2.5 mg albuterol sulfate nebulizer therapy with or without anticholinergic agent (ipratropium/tiotropium)
2. Patient is consented
3. Patient is randomized to receive either "Control Method" or "Study Method" first (see methods below)
4. The 1st morning after consent, the first study method is used
5. The 2nd morning after consent, the other study method is used
6. Study is over after the second study method is completed

Control Method:

1. Baseline patient data with spirometry is recorded including:

   Forced Vital Capacity (FVC), Forced Expiratory Volume in one second (FEV1),Forced Expiratory Ratio (FER), Peak Expiratory Flow (PEF), HR, Resting RR, Breath sounds, Pulse Oximetry (SpO2).
2. 2.5 mg albuterol sulfate is given with generic nebulizer for the 0700 treatment time. Anticholinergic agents such as ipratropium or tiotropium are given as ordered.
3. Follow-up patient data with spirometry is recorded at 15 minutes and 2 hours following the treatment.
4. Subsequent treatments that day are given as standard.

Study Method:

1. Baseline patient data with spirometry is recorded including:

   Forced Vital Capacity (FVC), Forced Expiratory Volume in one second (FEV1),Forced Expiratory Ratio (FER), Peak Expiratory Flow (PEF), Heart rate (HR), Resting respiratory rate (RR), Breath sounds, Pulse Oximetry (SpO2).
2. Albuterol sulfate (2.5 mg) is given via Aero Eclipse BAN with 0.5 ml of saline or 0.5 ml of ipratropium bromide (if ipratropium bromide is ordered).
3. Follow-up patient data with spirometry is recorded at 15 minutes and 2 hours following the treatment.
4. Subsequent treatments that day are given as ordered.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with orders for routine 2.5 mg albuterol sulfate nebulizer therapy ordered either Q4 or Q6 hours who consent to the study.

Exclusion Criteria:

* Adults with nebulizer therapy ordered more frequently than Q4 hours.
* Adults with nebulizer therapy ordered less frequently than Q6 hours.
* Pregnant patients are excluded.
* Adults with orders for albuterol sulfate > 2.5 mg.
* Adults in the ICU or Emergency Department.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity | 1
FEV1 | 1

CONTACTS AND LOCATIONS:
Overall Officials: John S. Emberger, BS, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Hospital, Newark, Delaware, United States